CLINICAL TRIAL: NCT01887262
Title: Control Of Fluid Balance Guided by Body Composition Monitoring in Patients on PeritoneAl dialySiS (COMPASS) Trial
Brief Title: Control Of Fluid Balance Guided by Body Composition Monitoring in Patients on PeritoneAl dialySiS
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Fresenius Medical Care Korea (Industry)
Responsible Party: Principal Investigator, Kook-Hwan Oh, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPASS
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Peritoneal Dialysis, Continuous Ambulatory
Keywords: fluid; edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Incident peritoneal dialysis (PD) patients who are randomly allocated to BCM-guided fluid management will receive BCM measurement every two months over 1-year period. The BCM results will be notified to the physicians and the participating subjects. Based on the BCM results along with the clinical information such as blood pressure, edema and weight, the physicians will prescribe PD fluid and diuretics, targeting within 1L of overhydration status. They will prescribe dietary education to the patient, if necessary.
  Interventions: Device: BCM-guided fluid management
- Control (Active Comparator): BCM will be measured at the beginning and end of the study, respectively. However, the BCM results will be blinded to the physicians and the control group. The physician will prescribe drugs, PD fluids, and dietary education to the patients based on the clinical information alone - such as blood pressure, edema and body weight.
  Interventions: Procedure: Fluid management based on the clinical information alone

INTERVENTIONS:
Device: BCM-guided fluid management
  Arms: Intervention
Procedure: Fluid management based on the clinical information alone
  Arms: Control

SUMMARY:
Bioimpedance-guided fluid management in peritoneal dialysis patients may provide better protection of residual renal function over 1 year period, compared with management guided by clinical information alone - such as blood pressure, body weight, and physician's physical examination.

ELIGIBILITY:
Inclusion Criteria:

* age bwten 20 and 75
* peritoneal dialysis > 4 weeks duration
* written consent
* daily urine output > 500 ml

Exclusion Criteria:

* subjects who are contraindicated to the bioimpedance measurement (pacemaker insertion state, defibrillator state, amputee, prosthesis, metal implants)
* pregnant women
* subjects who are expected to discontinue peritoneal dialysis with one year
* mixed dialysis modality (peritoneal + hemodialysis)
* hypoalbuminemic subjects (serum albumin < 3.3 g/dL)
* high blood pressure (> 160/100 mmHg despite antihypertensive medications)
* severe heart failure (NYHA FC III, or IV)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
delta GFR | baseline and 12th month
  change of glomerular filtration rate from baseline to the 12th month

SECONDARY OUTCOMES:
GFR | at 12th month
  glomerular filtration rate measured by urine collection, calculated by the mean of creatinine and urea clearance
time to anuria | over 12 months
  time to the anuric state (urine volume < 100cc/d)
echocardiographic parameters | 12 months period
  parameters obtained by echocardiographic measurements such as left ventracular mass index (LVMi), E/e' ratio, left vetricular end-diastolic volume (LVEDP), left ventracular ejection fraction (LVEF), left atrial volume indx (LAVI)
BP | 12th month
  systolic, diastolic blood pressure, pulse pressure
cardiovascular event | over 12 months
  fatal and nonfatal cardiovascular events - acute myocardial infarction (AMI), stroke, unstable angina, amputation, cardiovascular revascularization
BCM parameters | baseline and 12th month
  parameters measured by body composition monitoring (BCM), such as overhydration(OH), extracellular water (ECW), extracellular-to-intracellular water ratio (ECW/ICW)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

REFERENCES:
- [Background] Van Biesen W, Williams JD, Covic AC, Fan S, Claes K, Lichodziejewska-Niemierko M, Verger C, Steiger J, Schoder V, Wabel P, Gauly A, Himmele R; EuroBCM Study Group. Fluid status in peritoneal dialysis patients: the European Body Composition Monitoring (EuroBCM) study cohort. PLoS One. 2011 Feb 24;6(2):e17148. doi: 10.1371/journal.pone.0017148. PMID 21390320
- [Derived] Baek SH, Oh KH, Kim S, Kim DK, Joo KW, Oh YK, Han BG, Chang JH, Chung W, Kim YS, Na KY. Control of fluid balance guided by body composition monitoring in patients on peritoneal dialysis (COMPASS): study protocol for a randomized controlled trial. Trials. 2014 Nov 6;15:432. doi: 10.1186/1745-6215-15-432. PMID 25376940